CLINICAL TRIAL: NCT02482220
Title: Physical Activity and Energy Intake Control in Obese Adolescents: Effect of Exercise Programs of Various Intensities
Brief Title: Physical Activity Program and Energy Intake Control in Obese Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Blaise Pascal, Clermont-Ferrand (Other)
Responsible Party: Principal Investigator, THIVEL David, PhD, As/Pr, Research scientist, Université Blaise Pascal, Clermont-Ferrand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AU 1178
Record Dates: First submitted 2015-06-19; First posted 2015-06-26 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High intensity (Experimental): in this group, the participants will follow a high intensity physical activity program (High Intensity Interval exercise from 75 to 95% VO2max)
  Interventions: Behavioral: Physical activity intervention
- Moderate intensity (Experimental): in this group, the participants will follow a moderate intensity physical activity program (Intensity from 50 to 65% VO2max)
  Interventions: Behavioral: Physical activity intervention

INTERVENTIONS:
Behavioral: Physical activity intervention

SUMMARY:
Acute exercise of high intensity has been shown to induced nutritional adaptations in obese adolescents. Indeed, several studies have shown that about 30 minutes of intensive exercise (above 70% of the adolescents maximal aerobic capacities) can favor reduced-energy consumption at the following meal with no modification of their appetite feelings. Although it is suggested that chronic physical activity programs can induce energy intake modifications, this has never been clearly studied. The aim of this work is to compare different physical activity programs (low vs. high intensity programs) in terms of energy intake, appetite feelings and appetite-regulating hormones, in obese adolescents.

DETAILED DESCRIPTION:
After an first medical visit to ensure that the adolescents have the ability to complete the whole study, the participants will have to complete several clinical examinations:

* anthropometric measurements
* Body composition assessed by DXA
* Maximal aerobic test
* Blood samples (appetite-regulating hormones)
* daily energy intake assessment during a 24h intake exploration.

The adolescents recruited will then be randomly assigned to one of the two intervention groups:

- High Intensity program or moderate intensity program. Those two physical activity programs will last 4-months and will be composed of 3 to 4 exercise sessions per week. The High intensity program will consists in High intensity interval exercises starting at 70% of the adolescents' capacities at the beginning to end around 95%. The moderate intensity program will propose continuous exercises set between 50-65% VO2max.

No energy intake intervention will be performed.

By the end of the 4-months intervention, all the clinical examinations performed before the intervention will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 15 years old adolescents
* Obese according to international values for BMI
* Being registered to the national social security insurance
* no eating disorders
* no medications
* metabolic disorders

Exclusion Criteria:

* metabolic disorders
* food disorders
* physical disability

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
change in Energy intake in kcal is being assessed | energy intake will be assessed during 24h during the week before the intervention (T0) and the week after (T1)
  daily energy intake will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- AME2P Laboratory, Clermont-Ferrand, Auvergne, France